CLINICAL TRIAL: NCT04485507
Title: A Virtual Reality Intervention to Improve Attention in Heart Failure Patients
Brief Title: COgnitive Intervention to Restore Attention Using Nature Environment
Acronym: CORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Miyeon Jung, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1904370750
Record Dates: First submitted 2020-07-14; First posted 2020-07-24 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure; Cognitive Dysfunction
MeSH Terms: conditions — Heart Failure; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Two-group randomized controlled pilot study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature-VR (Experimental): Viewing 3D pictures of natural environments
  Interventions: Other: Nature-VR
- Urban-VR (Active Comparator): Viewing 3D pictures of urban environments
  Interventions: Other: Urban-VR

INTERVENTIONS:
Other: Nature-VR — Viewing 360 degree nature pictures delivered by a virtual reality headset for 10 minutes/day, 5 days/week for 4 weeks (total of 200 minutes).
  Arms: Nature-VR
Other: Urban-VR — Viewing 360 degree urban pictures delivered by a virtual reality headset for 10 minutes/day, 5 days/week for 4 weeks (total of 200 minutes).
  Arms: Urban-VR

SUMMARY:
Heart failure is a prevalent and serious public health concern with the growing aging population. Patients with heart failure often experience attention impairment that decreases their ability to perform self-care and diminishes their health-related quality of life. In past studies, 15 - 27% of heart failure patients had attention impairment. Attention is fundamental to human activities including self-care management of heart failure. However, cognitive interventions focusing on attention are scarce in heart failure literature. This study focuses on developing a novel cognitive intervention specifically targeting improved attention and testing its efficacy on improving attention, self-care, and health-related quality of life.

The investigators in this study are asking the following 3 questions: 1) does the newly developed cognitive intervention using immersive virtual reality technology (Nature-VR) improve attention compared with the control condition (Urban-VR)?; 2) does Nature-VR intervention improve HF self-care and health-related quality of life compared with Urban-VR control condition?; and 3) are selected biological factors associated with attention function in HF?

The virtual reality-based cognitive intervention (Nature-VR) can be an efficacious intervention for the patients to use and enjoy without burdening already reduced attention. This study has great potential to improve attention and prevent attention impairment, thereby leading to healthier lives among heart failure patients.

DETAILED DESCRIPTION:
Heart failure (HF) is a prevalent serious chronic illness that affects 6.5 million American. Among HF patients, prevalence of attention impairment is reported as 15-27%. Attention is fundamental to human activities including HF self-care. However, cognitive interventions focusing on attention are scarce in HF. The investigators developed a new cognitive intervention with immersive virtual reality technology and created a prototype of the virtual reality-based natural restorative environment intervention (Nature-VR). The prototype was feasible and showed larger effects in improving attention among 10 HF patients.

In this 2-group randomized controlled pilot study, specific aims are to: 1) examine preliminary efficacy of Nature-VR compared with Urban-VR on improving attention; 2) examine preliminary efficacy of Nature-VR compared with Urban-VR on HF self-care and health-related quality of life; and 3) explore possible biomarkers of attention in HF. This study is important and novel because this is the first intervention study targeting attention using virtual reality technology and investigating possible biomarkers associated with attention in HF patients.

ELIGIBILITY:
Inclusion Criteria:

* adults (> 21 years)
* diagnosed with chronic HF Stage C
* able to communicate in English

Exclusion Criteria:

* uncorrected visual impairment
* major neurological disease (e.g., Alzheimer disease, Parkinson's disease)
* major psychiatric disease (e.g., schizophrenia, bipolar disease)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Changes in attention - Multi-Source Interference Task | Baseline, 4 weeks, 8 weeks, 26 weeks, and 52 weeks
  Performances on the computerized cognitive test of Multi-Source Interference Task will be examined in terms of speed and accuracy. Participants are instructed to identify the target number, which is different than the other 3 numbers provided on the computer screen. There are two types of trials, congruent and incongruent. Congruent trials have a target number that is always matched its position on the button (e.g., 100, 020, or 223), in contrast, incongruent trials have the target number that is never matched with it position in the button (e.g., 010, 233, or 232). Faster response time and lower error rates indicate better attention.
Changes in attention - Digit Span Test | Baseline, 4 weeks, 8 weeks, 26 weeks, and 52 weeks
  Participants are instructed to remember the sequence of numbers the data collector told and repeat the numbers right after the instructor finished talking. This test has 2 subsets, Forward-repeat exactly the same sequence, and Backward-repeat the numbers in the backward from last to the first. More digits correctly repeated indicate better attention.
Changes in attention - Trail Making Test | Baseline, 4 weeks, 8 weeks, 26 weeks, and 52 weeks
  This traditional cognitive test of attention is a paper-pencil based measure and has 2 parts. Part A requires participants to connect a series of randomly arrayed, distinct circles numbered 1 to 25 in correct order as quickly as possible. Part B requires participants to connect a series of 25 circles numbered 1 to 13 randomly intermixed with letters from A to L, alternating between numbers and letters, and proceeding in ascending order (e.g., 1-A-2-B-3 and so on). Faster response time in seconds indicates better attention.
Changes in attention - Stroop Test | Baseline, 4 weeks, 8 weeks, 26 weeks, and 52 weeks
  Stroop Test is a color-word test measuring the ability to processe different visual features and ignore distractions. The test has 2 parts of reading letters of color names and colors of color names using 4 color names (i.e., red, blue, yellow, and green). Congruent trials have the same letters and colors of the color names (i.e., red in red color). Incongruent trials have different letters and colors of the color names (i.e., red in blue color). Faster response time and lower error rates indicate better attention.
Changes in attention - Attentional Function Index | Baseline, 4 weeks, 8 weeks, 26 weeks, and 52 weeks
  This self-reported questionnaire has 13 items on 0 to 10 response scales asking effectiveness in behaviors requiring attention. Higher scores indicate better subjective attention

SECONDARY OUTCOMES:
Changes in the Self-Care of Heart Failure Index (SCHFI) | Baseline, 4 weeks, 8 weeks, 26 weeks, and 52 weeks
  This self-reported questionnaire consists of 29 items divided into 3 scales measuring self-care maintenance, symptom perception, and self-care management. In addition, self-care confidence is measured by additional 10 items. Each scale is scored separately and standardized to achieve a possible score of 0 to 100. Higher scores indicate better self-care of HF.
Changes in Minnesota Living with Heart Failure Questionnaire (LHFQ) | Baseline, 4 weeks, 8 weeks, 26 weeks, and 52 weeks
  Minnesota Living with Heart Failure Questionnaire will be used to measure health-related quality of life. This self-report questionnaire consists of 21 items on which patients are asked to rate how their HF condition impacted their physical and emotional health. Lower scores indicate better HRQL.

OTHER OUTCOMES:
Changes in serum brain-derived neurotrophic factor levels (serum BDNF) | Baseline and 4 weeks
  Venipuncture will be performed to draw the blood by following Indiana University general laboratory safety guidelines. Changes in the serum BDNF levels (ng/ml) and its associations with attention will be examined.
BDNF gene | Baseline
  Venupucture will be performed to draw the blood for the possible genetic biomarker. The frequency of BDNF Val66Met genotype (e.g., rs6265) will be examined and attention will be examined by the genotype.
Apolipoprotein (APOE) gene | Baseline
  Venupucture will be performed to draw the blood for the possible genetic biomarker. The 3 common allele of APOE (i.e., e2, e3, and e4) will be examined. The frequency of APOE genotypes (e.g., rs7412, rs429358) will be examined and attention will be examined by the genotype.
Dopamine receptor gene | Baseline
  Venupucture will be performed to draw the blood for the possible genetic biomarker. Specifically, dopamine receptor gene 4 (e.g., 48 bp VNTR) polymorphism and its association with attention will be examined.
Dopamine transporter gene | Baseline
  Venupucture will be performed to draw the blood for the possible genetic biomarker. The dopamine transporter gene (DAT1) (e.g., rs28363170 - 40 bp VNTR) polymorphism and its association with attention will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Nursing, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided